CLINICAL TRIAL: NCT04565132
Title: High Definition Transcranial Direct Current Stimulation (HD-tDCS) for Chronic Tinnitus: Outcomes From a Prospective Longitudinal Large Cohort Study
Brief Title: HD-tDCS as a Treatment for Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDtDCS_extensive
Record Dates: First submitted 2020-08-12; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-08

CONDITIONS: Tinnitus, Subjective
Keywords: tinnitus; neuromodulation; non-invasive brain stimulation; transcranial direct current stimulation; large cohort; high-definition tDCS
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HD-tDCS (Experimental): Each patient received a total of six sessions of anodal HD-tDCS of right DLPFC.
  Interventions: Device: High Definition transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High Definition transcranial Direct Current Stimulation — 1x1 tDCS low-intensity stimulator and 4x1 multichannel stimulation adaptor (Soterix Medical Inc, New York, NY)

SUMMARY:
Transcranial Direct Current Stimulation (tDCS) aims to induce cortical plasticity by modulating the activity of brain structures. The broad stimulation pattern, which is one of the main limitations of tDCS, can be overcome with the recently developed technique called High-Definition tDCS (HD-TDCS). The objective of the current study is to investigate the effect of HD-tDCS on tinnitus in a large patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* chronic, subjective, non-pulsatile tinnitus
* met the criteria for HD-tDCS safety

Exclusion Criteria:

* a middle ear pathology
* another tinnitus treatment ongoing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Change in Tinnitus Functional Index (TFI) | Baseline (before intervention), immediately post intervention, 7 weeks follow-up
  Tinnitus severity self-report questionnaire, ranging from 0-100 with a higher score representing a more severe tinnitus

SECONDARY OUTCOMES:
Change in Visual Analogue scale (VAS) for tinnitus loudness | Baseline (before intervention), immediately post intervention, 7 weeks follow-up
  Visual analogue scale measuring tinnitus loudness from 0-100, with a higher score representing a louder tinnitus Visual analogue scale measuring tinnitus loudness from 0-100, with a higher score representing a louder tinnitus
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline (before intervention), immediately post intervention, 7 weeks follow-up
  Self-report questionnaire concerning anxiety and depression symptoms, ranging from 0-21 for each subscale. A result greater than 8 suggests the presence of a depression and/or anxiety disorder. Visual analogue scale measuring tinnitus loudness from 0-100, with a higher score representing a louder tinnitus
Change in Tinnitus Questionnaire (TQ) | Baseline (before intervention), immediately post intervention, 7 weeks follow-up
  Tinnitus severity self-report questionnaire, ranging from 0-84 with a higher score representing a more distressing tinnitus
Change in Hyperacusis Questionnaire (HQ) | Baseline (before intervention), immediately post intervention, 7 weeks follow-up
  Hyperacusis severity self-report questionnaire, ranging from 0-42 with a higher score representing a higher sensitivity to sounds. A score of 28 is the cut-off for auditory hypersensitivity.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacquemin L, Shekhawat GS, Van de Heyning P, Mertens G, Fransen E, Van Rompaey V, Topsakal V, Moyaert J, Beyers J, Gilles A. Effects of Electrical Stimulation in Tinnitus Patients: Conventional Versus High-Definition tDCS. Neurorehabil Neural Repair. 2018 Aug;32(8):714-723. doi: 10.1177/1545968318787916. Epub 2018 Jul 18. PMID 30019630
- [Background] Shekhawat GS, Sundram F, Bikson M, Truong D, De Ridder D, Stinear CM, Welch D, Searchfield GD. Intensity, Duration, and Location of High-Definition Transcranial Direct Current Stimulation for Tinnitus Relief. Neurorehabil Neural Repair. 2016 May;30(4):349-59. doi: 10.1177/1545968315595286. Epub 2015 Jul 15. PMID 26180052
- [Background] Shekhawat GS, Vanneste S. High-definition transcranial direct current stimulation of the dorsolateral prefrontal cortex for tinnitus modulation: a preliminary trial. J Neural Transm (Vienna). 2018 Feb;125(2):163-171. doi: 10.1007/s00702-017-1808-6. Epub 2017 Nov 10. PMID 29127483
- [Derived] Cardon E, Jacquemin L, Schecklmann M, Langguth B, Mertens G, Vanderveken OM, Lammers M, Van de Heyning P, Van Rompaey V, Gilles A. Random Forest Classification to Predict Response to High-Definition Transcranial Direct Current Stimulation for Tinnitus Relief: A Preliminary Feasibility Study. Ear Hear. 2022 Nov-Dec 01;43(6):1816-1823. doi: 10.1097/AUD.0000000000001246. Epub 2022 Jun 7. PMID 35666538